CLINICAL TRIAL: NCT04491292
Title: Psychosocial Impact of COVID-19 Pandemic on MD Anderson Workforce
Brief Title: Assessment of the Psychosocial Impact of the COVID-19 Pandemic on the MD Anderson Cancer Center Workforce
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0428; NCI-2020-04259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0428 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-28; First posted 2020-07-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Participants complete 2 online questionnaires over 10 minutes each at baseline and at 3 months after the pandemic ends.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the impact of the COVID-19 pandemic on the psychosocial health of employees of MD Anderson Cancer Center. Epidemics have been shown to promote psychological stress among medical staff in high risk areas, which may lead to mental health problems. Assessing how the pandemic is affecting employees may allow for more comprehensive actions to be taken to protect the mental health of employees.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess psychosocial and stress-related outcomes in employees at MD Anderson Cancer Center during and post the COVID-19 pandemic.

SECONDARY OBJECTIVE:

I. To identify demographic and occupational factors associated with COVID-19 related psychosocial and stress outcomes.

OUTLINE:

Participants complete 2 online questionnaires over 10 minutes each at baseline and at 3 months after the pandemic ends.

ELIGIBILITY:
Inclusion Criteria:

* MD Anderson employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in psychosocial outcomes | Baseline up to 3 months after the outbreak ends
  Will be assessed using the questions administered in the second part of the questionnaire, specifically, the 20 stress-related items and the Impact of Event Scale (IES). Summary statistics will be calculated for each of the individual 20 stress-related questions. The total distress score as well as the scores for the intrusion and avoidance subscales will be calculated and also summarized via descriptive statistics. Summary statistics will be calculated separately for data collected during the pandemic and at follow-up, as well as for change from pandemic to follow-up. Ninety-five percent confidence intervals will be calculated for the mean of the change scores.
Change in stress-related outcomes | Baseline up to 3 months after the outbreak ends
  Will be assessed using the questions administered in the second part of the questionnaire, specifically, the 20 stress-related items and the IES. Summary statistics will be calculated for each of the individual 20 stress-related questions. The total distress score as well as the scores for the intrusion and avoidance subscales will be calculated and also summarized via descriptive statistics. Summary statistics will be calculated separately for data collected during the pandemic and at follow-up, as well as for change from pandemic to follow-up. Ninety-five percent confidence intervals will be calculated for the mean of the change scores.

SECONDARY OUTCOMES:
Demographic and occupational factors associated psychological and stress-related outcomes | Up to 3 months
  Summary statistics will also be calculated for demographic variables as well as all other questionnaire items. Ninety-five percent confidence intervals will also be calculated for the mean change from the pandemic scores. Summary statistics will also be calculated for subgroups of interest, such as occupation, age, etc. Two-sided two-sample t-tests, analysis of variance or Pearson/Spearman correlation coefficients, as applicable, will be used to determine whether different subgroups are differentially impacted by, or whether different levels of demographics (such as age) or occupational factors (such as years of service at MD Anderson and number of hours worked per week) are associated with, the COVID-19-related stress, with the stress being measured by the total distress score calculated from the IES as well as by the intrusion and avoidance scores, separately during and after the pandemics.

CONTACTS AND LOCATIONS:
Overall Officials: Priya R Bhosale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org